CLINICAL TRIAL: NCT04206228
Title: Intravenous Iron Supplement for Iron Deficiency in Patients With Severe Aortic Stenosis: The IIISAS Trial
Brief Title: Intravenous Iron Supplement for Iron Deficiency in Patients With Severe Aortic Stenosis
Acronym: IIISAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars Gullestad, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-002037-11
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Severe Aortic Stenosis; Iron-deficiency
Keywords: Severe Aortic Stenosis; Iron-deficiency; Iron Isomaltoside; Exercise Capacity
MeSH Terms: conditions — Aortic Valve Stenosis; Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator): Active drug: Intravenous iron isomaltoside dissolved in 100 ml NaCl 0.9 %
  Interventions: Drug: Intravenous iron isomaltoside
- Placebo (Placebo Comparator): Placebo: Intravenous NaCl 0.9 % dissolved in 100 ml
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravenous iron isomaltoside — The active drug, iron isomaltoside, will be administered as a single, intravenous infusion of 20 mg/kg body weight (rounded off to the nearest 100 mg) dissolved in 100 ml NaCl as recommended by the drug manufacturer ("on-label" treatment), over 30 minutes only (1,67 ml/min).
  Other Names: Monofer®
  Arms: Active treatment
Drug: Placebo — The placebo will be prepared according to the randomisation code, and administered as a single intravenous infusion over 30 minutes only (1,67 ml/min).
  Other Names: Intravenous sodium chloride 0.9%
  Arms: Placebo

SUMMARY:
Iron deficiency is a prevalent nutritional deficiency and a common cause of anemia. Although iron deficiency is traditionally linked to anemia, iron deficiency is prevalent even in the absence of anaemia and in itself limits function and survival. Iron deficiency is a common feature of various chronic diseases, and up to 50% of patients with heart failure have iron deficiency. Iron deficiency is more prevalent the more advanced the disease is and occurs more frequently in women. Iron deficiency comprises absolute iron deficiency (usually defined as ferritin < 100 ng/ml) as well as functional iron deficiency, in which iron supply is inadequate to meet the demand for the production of red blood cells and other cellular functions despite normal or abundant body iron stores. Iron deficiency is associated with poor exercise capacity, lethargy and reduced quality of life. Results from our studies have shown that iron deficiency is prevalent in patients with aortic stenosis. Some of the symptoms associated with aortic stenosis, such as fatigue, reduced exercise capacity, dyspnoea and cognitive dysfunction, have traditionally been thought to be caused by the haemodynamic derangements precipitated by the valvular stenosis. However, similar symptoms can be brought about by iron deficiency, and the investigators hypothesize that intravenous iron supplement will improve exercise capacity, muscle strength, cognition, health-related quality of life and myocardial function in patients with severe aortic stenosis and iron deficiency. This is a phase 2, double blind, randomised, placebo-controlled trial. Participants will be randomised in a 1:1 fashion to receive a single intravenous dose of iron isomaltoside (50 patients) or matching placebo (50 patients). The study is designed to show superiority with regard to the primary endpoint in patients assigned to active treatment versus patients allocated to the placebo arm. The main goal is to evaluate the effect of a single dose of intravenous iron isomaltoside on exercise capacity after transcatheter aortic valve implantation in patients with severe aortic stenosis and iron deficiency. For this study, the investigators have defined as serum ferritin < 100 µg/l or ferritin between 100 and 300 µg/l in combination with a transferrin saturation < 20 %.

DETAILED DESCRIPTION:
Written informed consent must have been provided voluntarily by each subject before any study specific procedure is initiated.

A physical examination (including examination of heart, lungs, abdomen, neck and assessment of peripheral circulation and oedema) must be performed; vital signs (blood pressure, and heart rate); and height and weight must be recorded. A medical history must be obtained, and age; gender; New York Heart Association (NYHA) functional status; risk factors (hypertension, smoking, and diabetes); symptom duration, and concomitant disease must be recorded. All concomitant medication (incl. vitamins, herbal preparation and other "over-the-counter" drugs) used by the participant within 28 days of treatment start must be recorded in the CRF by generic name and dose. Blood samples will be obtained to determine haemoglobin; white blood cell count, platelet count; serum potassium; serum sodium; glucose, glycosylated haemoglobin; creatinine; ALT; bilirubin; albumin; INR; CRP; N-terminal pro-B-type natriuretic peptide; total cholesterol; ferritin; transferrin, serum iron and total iron binding capacity. Blood for efficacy analyses must be drawn and appropriately labelled and stored for later analysis. A 6 min walk test will be performed in accordance with current guidelines at baseline. The results of this test will be used for adjustment of the test-result six months after study drug infusion. The latter result, with adjustment for the baseline result, constitutes the primary endpoint of the IIISAS trial. Right and left hand grip strengths will be measured by a hand-held dynamometer. Body composition (weight, total water, total fat, percent fat, the ratio of extracellular water to intracellular water [measuring oedema], and visceral fat) will be measured at baseline and after 6 months with the InBody 770 body composition analyser. Self-reported, health-related quality of life will be gauged with the SF-36, EQ 5D 3L, EQ-VAS, HAD and the Kansas City Cardiomyopathy Questionnaires. Cognitive function will be assessed with the Cambridge Neuropsychological Test Automated Battery (CANTAB).

A physical examination, medical history, all concomitant medication, blood samples, 6 min walk test, right and left hand grip strengths, body composition, and self-reported, health-related quality of life as well as cognitive function will be conducted again on average approximately 3 months after study drug administration, and it is designed to assess initial efficacy and safety. This will be conducted again 3 months after transcatheter aortic valve implantation (TAVI).

Patients will be followed for the first year after the TAVI procedure for safety assessment, including MACE, and all-cause mortality. At 12 months after that TAVI procedure, approximately 15 months after study drug infusion, a visit to Oslo University hospital, the local hospital or a telephone interview will be performed to assess NYHA functional class, adverse events and clinical events.

Patients may be discontinued from study treatment and assessments at any time. Specific reasons for discontinuing patient follow-up are:

* Voluntary discontinuation: participating patients are free to discontinue his/her participation in the study at any point in time, without prejudice to further treatment.
* Major protocol deviation
* Incorrect randomisation, i.e. the patient does not meet the required inclusion/exclusion criteria for the study
* Patient lost to follow-up
* Patient's non-compliance to study treatment and/or procedures

Patient withdrawal must be documented in the CRF as well as in hospital records. If possible, a final assessment should be obtained (end of study visit). The reason for discontinuation is recorded. The investigator is obliged to follow up any significant adverse events until the outcome either is recovered or resolved, recovering/resolving, not recovered/not resolved, recovered/resolved with sequelae, fatal or unknown. Patients who withdraw will be included in the intention-to treat analysis.

The whole trial may be discontinued at the discretion of the primary investigator or the sponsor in the event of any of the following:

* Occurrence of AEs unknown to date in respect of their nature, severity and duration
* Medical or ethical reasons affecting the continued performance of the trial
* Difficulties in the recruitment of patients
* Cancellation of drug development The sponsor and principal investigator will inform all investigators, the relevant Competent Authorities and Ethics Committees of the termination of the trial along with the reasons for such action. If the study is terminated early on grounds of safety, the Competent Authorities and Ethics Committees will be informed within 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Aortic stenosis patients with peak flow velocity (>3.5 m/s) scheduled for aortic valve replacement with TAVI
* Iron deficiency defined as serum ferritin < 100 µg/l or ferritin between 100 and 300 µg/l in combination with a transferrin saturation < 20 %.
* Age > 18 years.
* Signed informed consent and expected compliance with protocol.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

* Anaemia (Haemoglobin < 100 mg/l)
* Haemochromatosis
* Haemosiderosis
* Porphyria cutanea tarda
* Blood dyscrasias or any disorders causing haemolysis or unstable red blood cells
* Decompensated liver disease (Child-Pugh score 7 or higher)
* End-stage renal failure, i.e. eGFR < 15 ml/min or on renal replacement therapy
* Planned major surgery within 6 months
* On erythropoietin analogues
* Known sensitivity or intolerance to iron isomaltoside or other parenteral iron preparations
* Intravenous iron supplement within 6 months prior to inclusion
* A clear indication for intravenous iron supplement
* On oral iron substitution (unless the subject agrees to stop treatment prior to randomisation)
* Alcohol or drug abuse within 3 months of informed consent that would interfere with trial participation or any ongoing condition leading to decreased compliance with study procedures or study drug intake
* Intake of an investigational drug in another trial within 30 days prior to intake of study medication in this trial or participating in another trial involving an investigational drug and/or follow-up
* Failure to obtain written informed consent
* Inability to walk at least 100 meters over 6 minutes
* Women of child-bearing potential (1)

  1. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Menopause is defined as 12 months continuous amenorrhea without an alternative medical cause in a female ≥ 55 years old or 12 months of spontaneous and continuous amenorrhea with a follicle stimulating hormone (FSH) level > 40 IU/L (or according to the definition of "postmenopausal range" for the laboratory involved) in a female < 55 years old unless the subject has undergone bilateral oophorectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Submaximal Exercise Test | 6 months
  The baseline-adjusted distance walked on a 6 min walk test performed 6 months after the trial intervention.

SECONDARY OUTCOMES:
Iron deficiency | 6 months
  Iron deficiency defined as serum ferritin < 100 µg/l or ferritin between 100 and 300 µg/l in combination with a transferrin saturation < 20 %.
Muscle strength | 6 months
  Grip strength will be measure using a hand-held dynamometer (hand-grip device).
The 36-item short health survey questionnaire (SF-36) | 6 months
  The SF-36 Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
The 3-level version of EQ-5D (EQ-5D-3L) questionnaire | 6 months
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
EuroQol-visual analogue scales (EQ-VAS) | 6 months
  EQ-VAS is an instrument to measure overall health on a vertical visual analogue scale, ranging from "worst possible" (zero) to "best possible" (100)health.
Hospital anxiety and depression scale (HADS) | 6 months
  HADS is a fourteen item scale used to determine the levels of anxiety and depression that a person is experiencing. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
The Kansas City Cardiomyopathy Questionnaire (KCCQ) | 6 months
  KCCQ is a 23-item, self administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The responses are categorized under 3 subscales (symptom burden, physical limitation and quality of life) with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms.
Cambridge Neuropsychological Test Automated Battery (CANTAB) (www.cambridgecognition.com) | 6 months
  CANTAB (www.cambridgecognition.com) is a computer-based cognitive assessment system consisting of a battery of seven neuropsychological tests, administered to subjects using a touch screen computer. Automatic scoring, adjusted for age, gender and education level.
N-terminal pro-B-type natriuretic peptide (NT-proBNP) | 6 months
  NT-proBNP is measured as a simple blood test and used as diagnostic biomarker for heart failure and cardiac dysfunction in clinical medicine.
Cardiac troponin T (TnT) | 6 months
  TnT is measured as a simple blood test and used as a standard biomarker of myocardial injury.
Number of adverse events (AE) | 6 months
  The standard time period for collecting and recording AE and SAEs will begin at the start of study treatment and the mandatory reporting of new AEs ends after the end-of-study visit 6 months after study drug infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Gullestad, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bardan S, Kvaslerud AB, Andresen K, Klove SF, Edvardsen T, Gullestad L, Broch K. Intravenous ferric derisomaltose in iron-deficient patients undergoing transcatheter aortic valve implantation due to severe aortic stenosis: study protocol of the randomised controlled IIISAS trial. BMJ Open. 2022 Sep 2;12(9):e059546. doi: 10.1136/bmjopen-2021-059546. PMID 36691165
- [Derived] Kvaslerud AB, Bardan S, Andresen K, Klove SF, Fagerland MW, Edvardsen T, Gullestad L, Broch K. Intravenous iron supplement for iron deficiency in patients with severe aortic stenosis scheduled for transcatheter aortic valve implantation: results of the IIISAS randomised trial. Eur J Heart Fail. 2022 Jul;24(7):1269-1279. doi: 10.1002/ejhf.2557. Epub 2022 Jun 3. PMID 35579454